CLINICAL TRIAL: NCT04939077
Title: Treatment of Heart Failure Using Human Umbilical Cord Mesenchymal Stem Cells(hUC-MSC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MR-31-20-000323
Record Dates: First submitted 2020-12-03; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Myocardial Ischemia; Ventricular Dysfunction, Left
Keywords: Human Umbilical Cord Mesenchymal Stem Cells; Heart Failure
MeSH Terms: conditions — Myocardial Ischemia; Ventricular Dysfunction, Left; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CABG with hUC-MSC treatment group (Experimental): In the CABG with hUC-MSC treatment group, 1×10^7 human umbilical cord Mesenchymal Stem Cells were injected to the edge of the myocardial infarction area at 20 points at the same time in CABG.
  Interventions: Biological: Allogeneic Human Umbilical Cord Mesenchymal Stem Cells
- CABG group (No Intervention): CABG was performed under general anesthesia.

INTERVENTIONS:
Biological: Allogeneic Human Umbilical Cord Mesenchymal Stem Cells — In CABG with hUC-MSC treatment group, 1×10^7 Human Umbilical Cord Mesenchymal Stem Cells were injected at the edge of the myocardial infarction area at 20 points at the same time in CABG
  Arms: CABG with hUC-MSC treatment group

SUMMARY:
This study is an exploratory clinical study to observe the improvement of heart function before and after the treatment by human umbilical cord mesenchymal stem cells, and the purpose is to evaluate the safety and effectiveness of human umbilical cord mesenchymal stem cells in the treatment of heart failure. The study is a randomized parallel controlled study. Patients receive a review of which main content includes symptom improvement, cardiac function improvement, and adverse events.

DETAILED DESCRIPTION:
This study is an exploratory clinical study to observe the improvement of heart function before and after the treatment by human umbilical cord mesenchymal stem cells, and the purpose is to evaluate the safety and effectiveness of human umbilical cord mesenchymal stem cells in the treatment of heart failure. The study is a randomized parallel controlled study. The research process is as follows: 1. Twenty eligible patients with ischemic heart disease were recruited, fully informed, and signed a consent form, and randomly divided into CABG group (n=10) or CABG + stem cell treatment group (n=10); 2. CABG was performed under general anesthesia in both groups. In the cell therapy group, 1×10^7 human umbilical cord Mesenchymal Stem Cells were injected to the edge of the myocardial infarction area at 20 points at the same time in CABG; 3. Use vasoactive drugs and antibiotics to prevent infection one week after surgery. After the operation, before discharge, 1 month, 3 months, 6 months, 12 months after discharge, and once a year thereafter, until the death of the patient. Patients receive a review of which main content includes symptom improvement, cardiac function improvement, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* The patients with coronary heart disease, the effect of drug treatment is not good, and the clinical manifestations of left ventricular insufficiency occur, EF<40%;
* Coronary angiography confirmed that there is a chronic occlusive disease of the coronary artery, which is manifested as severe stenosis of single or multiple coronary vessels (≥75%), or even complete occlusion;
* After the doctor explained the treatment process and possible toxic and side effects, he was willing to treat and agreed to cooperate in the observation of the efficacy. But patients can withdraw from clinical trials and long-term follow-up observation at any time and unconditionally;
* The patient has no mental illness and language dysfunction and can fully understand the treatment method.

Exclusion Criteria:

* Does not meet the above selection criteria;
* Unable to sign the informed consent form, unable to comply with the agreed timetable of this study;
* There are reasons to suspect that the patient was forced to join the trial;
* Acute left ventricular insufficiency, cardiogenic shock;
* The patient has any infectious diseases (including bacterial and viral infections);
* Others who are clinically considered unsuitable for this treatment.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-27 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | Day 0, Day 30, Day 90, Day 180, Day 360, Day 720
  The change in Left ventricular ejection fraction (LVEF) % after the operation
Left ventricular end diastolic volume | Day 0, Day 30, Day 90, Day 180, Day 360, Day 720
  The change in Left ventricular end diastolic volume (LVEDV) ml after the operation
Left ventricular end systolic volume | Day 0, Day 30, Day 90, Day 180, Day 360, Day 720
  The change in Left ventricular end systolic volume (LVESV) ml after the operation
Stroke volume | Day 0, Day 30, Day 90, Day 180, Day 360, Day 720
  The change in Stroke volume (SV) ml after the operation
Left ventricular apex four-chamber end systolic diameter | Day 0, Day 30, Day 90, Day 180, Day 360, Day 720
  The change in Left ventricular apex four-chamber end systolic diameter (LVESD) mm after the operation
6 minutes walking distance | Day 0, Day 30, Day 90, Day 180, Day 360, Day 720
  The change in 6 minutes walking distance m after the operation

SECONDARY OUTCOMES:
THE WORLD HEALTH ORGANIZATION QUALITY OF LIFE (WHOQOL) -BREF | Day 0, Day 30, Day 90, Day 180, Day 360, Day 720
  The change in THE WORLD HEALTH ORGANIZATION QUALITY OF LIFE (WHOQOL) -BREF after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Zhongmin Liu, Doctor, Principal Investigator — Shanghai East Hospital, Shanghai Tongji University
Locations (1):
- Shanghai East Hospital, Shanghai Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided